CLINICAL TRIAL: NCT06179394
Title: Evaluation of Cognitive Dysfunction and Psychiatric Comorbidities in Patients With Wilson Disease
Brief Title: Evaluation of Cognitive Dysfunction and Psychiatric Comorbidities
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mustafa Ahmed Sedky Abdallah, doctor, Assiut University
Other Study IDs: Wilson disease
Record Dates: First submitted 2023-12-12; First posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Wilson Disease
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary objective

* Collection of patients with wilson disease either presented with neurological or hepatic symptoms
* Assessment of psychiatric and cognitive disorders in both groups by using specific scales Secondary objective
* correlation of MRI brain findings with cognitive & psychiatric symptoms found in the patients ,if possible.

DETAILED DESCRIPTION:
Wilson's disease is an autosomal recessive disorder of copper metabolism caused by ATP7B mutations. Originally described as hepatolenticular degeneration, it classically presents with the combination of liver disease and a movement disorder during adolescence or early adulthood, albeit with a highly variable phenotype. Up to 60% of patients have neurological or psychiatric symptoms at onset, and are referred to as having neurological presentations (1). Chelating agents are used to 'de-copper' patients but neurological outcomes are unpredictable; symptoms usually improve however, a minority have persistent or progressive neurological disability (2, 3).

It is clinically relevant that the severity of neurologic symptoms commonly fluctuates, sometimes during the same day. Symptoms may be exacerbated by stress, concurrent illnesses, or medications (4). WD has been associated with multiple cognitive, emotional, or psychiatric disorders, which may occur at any stage of disease (5 ). The first psychiatric manifestation of WD could occur in childhood and appear as a decline in school performance, inappropriate behavior or impulsiveness(6). It is common to observe classic psychiatric syndromes in later early adulthood, including behavioral and personality changes, anxiety, depression, manic and hypomanic syndrome, cognitive deficits (7-10). personality and behavioral disorder due to brain disease, damage and dysfunction' (11).The BG are a structure capable of generating diverse psychiatric syndromes under dysfunctional conditions. Cognitive impairment in WD patients with neuropsychiatric presentation is well described (12) and probably related to the cerebral lesions detected by MRI (13). WD patients will firstly experience prospective memory related to the planning or goal-making of daily activities (14), which is associated with gray matter loss in the basal ganglia and structural changes in frontal and occipital whiter matter (15).

ELIGIBILITY:
Inclusion Criteria:

* age 8-70, both sexes, diagnosed as Wilson disease.

Exclusion Criteria:

* • Patients with neurological symptoms due to neurological disease other than Wilson disease such as patients with cerebrovascular stroke or Parkinson disease, ……

  * Patients with hepatic encephalopathy or severe neurological impairments (disabling dysarthria, tremor or dystonia) or severe psychiatric disorders incompatible with neuropsychological examination
  * Patients with liver transplant

Ages: 8 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: all pt fulfilling inclusion criteria will including in my study except that we exculded .
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-12-15 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
correlation | base line
  • correlation of MRI brain findings with cognitive & psychiatric symptoms found in the patients